CLINICAL TRIAL: NCT05050916
Title: The Investigation of Vitamin D and Menstrual Cycles Trial: A Phase II Clinical Trial
Brief Title: The Investigation of Vitamin D and Menstrual Cycles Trial, the inVitD Trial: A Phase II Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10000476; 000476-E (Other: NIH IRB)
Record Dates: First submitted 2021-09-18; First posted 2021-09-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-07-09

CONDITIONS: Reproductive Issues
Keywords: reproductive; Health; Female; Hormones; period
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1/High Dose Vitamin D (Experimental): Deficient participants will be assigned to the Endocrine Society recommendation for deficiency, 50,000 IU/week.
  Interventions: Dietary Supplement: Vitamin D
- 2/Placebo (Placebo Comparator): Participants with sufficient levels of vitamin D will receive placebo instead of Vitamin D supplementation.
  Interventions: Other: Placebo
- 3/Low Dose Vitamin D (Experimental): Early in the study, deficient participants were randomized to either the U.S. recommended daily allowance, 4200 IU/week or the high dose vitamin D arm. The low dose arm was discontinued mid-way through the trial and all deficient participants were assigned to the high dose arm.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — The High Dose Vitamin D arm will receive 50,000 IU/week of cholecalciferol. The Low Dose Vitamin D arm will receive 4,200 IU/week of cholecalciferol
  Arms: 1/High Dose Vitamin D; 3/Low Dose Vitamin D
Other: Placebo — Cellulose capsule
  Arms: 2/Placebo

SUMMARY:
Background:

About 1.5 million U.S. women of reproductive age are estimated to be infertile. Many more have difficulty getting pregnant. Menstrual cycles are an indicator of a woman's general health. Menstrual cycle changes may predict difficulties in getting pregnant. Researchers want to see what role vitamin D may play in menstrual cycle health.

Objective:

To examine the effect of vitamin D supplementation on the hormones that come from the brain and the ovary during a menstrual cycle.

Eligibility:

Women aged 19-40 who have spontaneous menstrual cycles (are not taking any hormones) less than 50 days in length.

Design:

Participants will fill out a screening survey about their demographics and health history. It will take 5-10 minutes to complete.

Participants will have 3 study visits. Participants who have low vitamin D and move to Phase 2 will receive 50000 IU//week of vitamin D supplement. Participants who do not have low vitamin D will receive placebo. If they have low vitamin D, they will not get the placebo. They will take the capsules by mouth, once per week, for 3 menstrual cycles (or about 90 days).

Participants will have physical exams. Their height, weight, body fat percentage, blood pressure, and waist-hip ratio will be measured. They will give blood samples. They will self-administer vaginal and oral swabs.

Participants will keep a daily menstrual diary. They will do daily home ovulation testing. They will collect urine at home. Some women may collect menstrual blood at home.

Participants will fill out an online survey. It will ask about their health, diet, and physical activity; birth control use; pregnancy history; menstrual cycle; smoking and drinking habits; education; and occupation. It will take 20-30 minutes to complete.

Participation will last for four menstrual cycles (about 4 months).

DETAILED DESCRIPTION:
Study Description:

This Phase II clinical trial translates both animal studies and human observational research into public health relevant research. We will investigate vitamin D's influence on the hypothalamic-pituitary-ovarian axis by careful evaluation of hormonal and ovulatory menstrual cycle changes that occur with vitamin D supplementation. Vitamin D supplementation may be a low-cost intervention that improves menstrual cycle function and fertility.

After recruitment, there will be two phases to this study: Phase 1 will follow all women for at least one menstrual cycle prior to supplementation, the pre-supplementation cycle. During Phase 1, blood will be drawn and assayed for 25-hydroxyvitamin D (25OHD). If their level is less than 20 ng/ml, they will be invited to participate in Phase 2. A small sample of participants with a level >= 20 ng/ml will also be invited to participate in Phase 2, to maintain participant blinding. Participation ends for the remaining participants whose level is 20 ng/ml or higher. During Phase 2, those with low vitamin D receive a blinded dose of 50,000 IU/week of vitamin D supplementation. The small group of sufficient participants will receive a placebo. Participants will not be told what their 25OHD level was. Women will be followed for three more menstrual cycles. In the pre-supplementation cycle and in the last supplemented cycle, women will collect daily urine specimens. Hormone levels will be compared between the pre-supplementation and supplemented cycles as the primary analysis. A secondary analysis will compare the supplemented cycles in those who received 50,000 IU and those who received placebo.

The original design of this trial included a low-dose (4,200 IU) vitamin D supplementation arm. At entry into Phase 2, participants were randomized to receive the 4,200 IU/week vitamin D supplement or 50,000 IU/week vitamin D supplement in a 2:3 ratio. The low-dose arm of the trial has been discontinued for cost and efficiency purposes. As of 12/13/22, 16 participants were randomized to receive the low-dose vitamin D supplement. On approval of the current document, this information will be updated to reflect the final count of participants who received the low-dose vitamin D supplement and the specific date at which the low-dose arm was discontinued via a future amendment. Study data for those who received the low-dose vitamin D supplement will be retained for research and analysis. Specific analyses, biospecimen use, and statistical comparisons will not differ from those described below for the participants who receive the 50,000 IU vitamin D supplement or the placebo. All data handling and security procedures described in this document equivalently apply to data collected from participants receiving the low-dose vitamin D supplement.

The primary aim of this trial will test the following hypotheses by comparing vitamin D supplemented cycles to the pre-supplementation cycles, within-woman: (1) Mid-luteal progesterone is higher in vitamin D supplemented cycles; (2) Rate of estrogen rise is higher in vitamin D supplemented cycles; (3) Pre-ovulatory luteinizing hormone (LH) is higher in vitamin D supplemented cycles.

Objectives:

Primary objective:

-To examine the effect of vitamin D supplementation on hypothalamic-pituitary-ovarian axis hormones. We will evaluate the extent to which vitamin D supplementation:

* Increases urinary mid-luteal progesterone (an indicator of healthy, fertile follicle development)
* Increases the rate of rise in urinary follicular phase estrogen (an indicator of follicular development)
* Increases urinary pre-ovulatory LH (an indicator of healthy ovarian-hypothalamic interaction)

Secondary objectives:

* Determine the impact of vitamin D supplementation in reproductive-aged women by assaying the metabolome before and after vitamin D supplementation
* To quantify the increase in 25OHD and the fraction who achieve a level of 40 ng/ml after 1.5 and 3 months of supplementation, in response to 50,000 IU/week of vitamin D.
* To examine the effects of vitamin D supplementation on endometrial stromal cell decidualization

Tertiary/Exploratory objectives:

* To examine the change in whole blood metals levels in response to vitamin D supplementation.
* To examine the change in vaginal or oral microbiome in response to vitamin D supplementation.
* To investigate the extent to which vitamin D reduces the incidence of

  --delayed ovulation (follicular phase >20 days), 2) short luteal phase (<=10 days), and 3) long cycles (>34 days)
* To investigate the association between 25OHD levels, sleep measures, physical activity, exposure to white/red/green/blue light, and hypothalamic-pituitary-ovarian axis hormones.

Endpoints:

Primary Endpoint: Mid-luteal progesterone, follicular estrogen, preovulatory LH

Secondary Endpoints: Untargeted metabolomics, 25OHD, endometrial stromal cell function,

Tertiary Endpoints: metals, microbiome, ovulation, menstrual cycle length, sleep

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Having natural, spontaneous menstrual cycles (no hormonal therapy) less than 50 days in length.
* Aged 19-40 years
* Ability to take a vitamin D capsule and willing to adhere to the weekly regimen
* If sexually active, use of a non-hormonal contraceptive method.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* No menstrual period in the last 50 days, or, a typical menstrual cycle length <16 or >49 days.
* Use of a vitamin D supplement for more than one month and on more than 15 days out of each month. Volunteers will be asked to check their supplement label for vitamin D content.
* Unwilling to abstain from taking non-study vitamin D supplements during the study or if already taking a medically-advised vitamin D supplement.
* Use of a calcium supplement (including certain antacids) and unwilling to abstain from taking a calcium supplement during the study.
* Known polycystic ovarian syndrome
* Depo-provera use in the previous 12 months
* Current use of any hormones, including birth control
* Current use of a hormonal intrauterine device (IUD)
* Current pregnancy or lactation, trying to become pregnant, or planning to try in the next four menstrual cycles or 5 months.
* History of seizure disorders
* Celiac disease
* Crohn s Disease
* Body mass index >35
* Aged <19 or > 40 years
* Presence of known contraindications for vitamin D supplementation, history of any of the following: calcium disorder or hypercalcemia, tuberculosis or granulomatous disease, metastatic bone disease, sarcoidosis, Williams syndrome, kidney disease (kidney stones, renal failure or dialysis, lupus nephritis)
* Known liver disease (cirrhosis)
* History of cancer other than skin cancer.
* History of anorexia nervosa, bulimia or an eating disorder
* Use within the past 60 days, of exogenous hormones
* Type 1 or Type 2 diabetes
* Known heart disease
* Gastric bypass surgery
* Unwilling or unable to complete study activities, e.g. collect daily urine specimens, have blood drawn, complete daily diaries, attend in person study visits

  25. Non-English speaking
* Due to the complexity of daily/weekly diaries, testing and procedurerequirements, all consents, instructions and questionnaires are provided in English. Therefore, all participants must be able to able to read and speak English.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
To examine the effect of vitamin D supplementation on hypothalamic-pituitary-ovarian axis hormones. | 60 months
  We will evaluate the extent to which vitamin D supplementation: 1) Increases urinary mid-luteal progesterone (an indicator of healthy, fertile follicle development) 2) Increases the rate of rise in urinary follicular phase estrogen (an indicator of follicular development) 3) Increases urinary pre-ovulatory LH (an indicator of healthy ovarian-hypothalamic interaction)

SECONDARY OUTCOMES:
To quantify the increase in 25OHD and the fraction who achieve a level of 40 ng/ml after 1.5 and 3 months of supplementation, in response to 50,000 IU/week of vitamin D. | 60 months
  25OHD
To investigate the effect of vitamin D supplementation on the microbiome | 60 months
  Untargeted microbiome profiling
To investigate the effect of vitamin D supplementation on endometrial stromal cell function. | 60 months
  Endometrial stromal cells isolated from menstrual effluent.
To examine the change in whole blood metals levels in response to vitamin D supplementation. | 60 months
  Whole blood lead
Determine the impact of Vitamin D supplementation in reproductive-aged women by assaying the metabolome before and after vitamin D supplementation. | 60 months
  Untargeted metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Z Jukic, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Metz CN, Chatterjee PK, Hyman N, Busch S, Tarasenko SA, Hoofnagle AN, Gregersen PK, Steiner AZ, Jukic AMZ. Leveraging menstrual effluent (ME) to investigate vitamin D and human decidualization, a potential link with fertility. J Clin Endocrinol Metab. 2026 Jan 5:dgaf708. doi: 10.1210/clinem/dgaf708. Online ahead of print. PMID 41492807
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000476-E.html